CLINICAL TRIAL: NCT06326489
Title: Evaluating the Efficacy and Quality of Life Impact of Transitioning to Advanced Hybrid Closed-Loop Insulin Pump Therapy in Romanian Children With Type 1 Diabetes Mellitus
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: ELIAS Emergency University Hospital (Other)
Responsible Party: Principal Investigator, Ioacara Sorin, Assoc. Prof. Dr., ELIAS Emergency University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105122023-1/05.12.2023; ERP-2023-13520 (Other Grant/Funding Number: Medtronic)
Record Dates: First submitted 2024-03-17; First posted 2024-03-22 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: HbA1c; insulin pumps; closed-loop
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: The study will include 30 children with type 1 diabetes aged seven years and older who use a predictive low glucose suspend insulin pump (740G). Patients eligible for the study will receive a 780G insulin pump for three months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 780G (Experimental): Patients in this arm will receive a 780G for three months.
  Interventions: Device: Switching to the Medtronic 780G insulin pump

INTERVENTIONS:
Device: Switching to the Medtronic 780G insulin pump — Patients using a Medtronic 740G insulin pump will receive the 780G model for three months

SUMMARY:
The proposed study aims to demonstrate the potential benefits of transitioning T1DM children from predictive low glucose suspend insulin pump therapy to advanced hybrid closed-loop insulin pump therapy in Romania. Primary Outcome: Variations in HbA1c between baseline visit (V1 - 740G) and assessment visit following three months of 780G insulin pump therapy (V2 - 780G).

Secondary Outcomes: changes in insulin requirements, time in range (TIR) levels, time below range (TBR), coefficient of variation (CV), frequency of severe hypoglycemic and hyperglycemic events requiring hospitalization, and PedsQL SF15 questionnaire scores.

ELIGIBILITY:
Inclusion Criteria:

* Age 7 years or older at baseline
* Diagnosis of type 1 diabetes
* Current use of a predictive low glucose suspend insulin pump (740G)
* At least 30% of subjects must have an HbA1c > 7,5% (58 mmol/mol)

Exclusion Criteria:

* Age < 7 years or ≥ 18 years at baseline
* Diabetes duration < 1 year at baseline
* HbA1c ≤ 7% (53 mmol/mol)
* Not meeting the Romanian national standards for closed-loop insulin pump therapy
* Other criteria deemed inappropriate by the principal investigator (to be documented)

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Variations in HbA1c | Three months
  Variations in HbA1c between baseline visit (V1 - 740G) and assessment visit following three months of 780G insulin pump therapy (V2 - 780G)

SECONDARY OUTCOMES:
changes in insulin requirements | Three months
  changes in insulin requirements between baseline visit (V1 - 740G) and assessment visit following three months of 780G insulin pump therapy (V2 - 780G)
changes in time in range (TIR) levels | Three months
  changes in time in range (TIR) levels between baseline visit (V1 - 740G) and assessment visit following three months of 780G insulin pump therapy (V2 - 780G)
changes in time below range (TBR) | Three months
  changes in time below range (TBR) between baseline visit (V1 - 740G) and assessment visit following three months of 780G insulin pump therapy (V2 - 780G)
changes in coefficient of variation (CV) | Three months
  changes in coefficient of variation (CV) between baseline visit (V1 - 740G) and assessment visit following three months of 780G insulin pump therapy (V2 - 780G)
changes in frequency of severe hypoglycemic and hyperglycemic events requiring hospitalization | Three months
  changes in frequency of severe hypoglycemic and hyperglycemic events requiring hospitalization between baseline visit (V1 - 740G) and assessment visit following three months of 780G insulin pump therapy (V2 - 780G)
changes in The Pediatric Quality of Life Inventory™ 4.0 Short Form 15 Generic Core Scales questionnaire scores | Three months
  changes in The Pediatric Quality of Life Inventory™ 4.0 Short Form 15 Generic Core Scales questionnaire scores between baseline visit (V1 - 740G) and assessment visit following three months of 780G insulin pump therapy (V2 - 780G). Scores are transformed on a scale from 0 to 100. Higher scores = Better Quality of Life

CONTACTS AND LOCATIONS:
Locations (1):
- Elias University Emergency Hospital, Bucharest, Sector 1, Romania

IPD SHARING:
Plan to Share IPD: No